CLINICAL TRIAL: NCT01192451
Title: Prospective Cohort of Patients With Chronic Obstructive Pulmonary Disease (COPD) Undergoing Domiciliary Noninvasive Positive Pressure Ventilation
Brief Title: Prospective Cohort of Respiratory Insufficiency Outcome
Acronym: RIO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Professeur jean-François Timsit, Grenoble university hospital
Other Study IDs: 08SC01
Record Dates: First submitted 2010-08-30; First posted 2010-09-01 (Estimated); Last update posted 2010-09-13 (Estimated); Status verified 2010-09

CONDITIONS: COPD; Non Invasive Ventilation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The Respiratory Insufficiency Outcome (RIO) project consists in a french multicenter prospective cohort of patients with chronic obstructive pulmonary disease (COPD) undergoing domiciliary noninvasive positive pressure ventilation.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of COPD
* domiciliary noninvasive ventilation

Exclusion Criteria:

* noninvasive ventilation set up for a neuromuscular disease

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: COPD patients undergoing domiciliary noninvasive ventilation
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2008-12

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - University Hospital, Grenoble
  - Hopital de La Croix Rousse, Lyon
  - Hopital de La Pitie Salpetriere, Paris
  - Hopital Nord, Saint-Etienne

REFERENCES:
- [Derived] Borel JC, Pepin JL, Pison C, Vesin A, Gonzalez-Bermejo J, Court-Fortune I, Timsit JF. Long-term adherence with non-invasive ventilation improves prognosis in obese COPD patients. Respirology. 2014 Aug;19(6):857-65. doi: 10.1111/resp.12327. Epub 2014 Jun 9. PMID 24912564